CLINICAL TRIAL: NCT01194622
Title: Single Dose Pharmacokinetics of Intranasal Fluticasone Delivered by a Fixed Combination With Azelastine (MP29 02) in Comparison to Two Different Fluticasone Nasal Sprays Single-centre, Randomised, Open-label, Three-period, Six-sequence Cross-over Trial (William's Design)
Brief Title: Single Dose Pharmacokinetics of Intranasal Fluticasone Delivered by a Fixed Combination With Azelastine (MP29 02) in Comparison to Two Different Fluticasone Nasal Sprays
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MEDA Pharma GmbH & Co. KG (Industry)
Collaborators: ClinResearch, GmbH (Other); Prolytic GmbH (Industry); pharm-analyt GmbH (Unknown)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: X-03065-3282; 2010-019557-18 (EudraCT Number)
Record Dates: First submitted 2010-09-02; First posted 2010-09-03 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2016-04

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — azelastine; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Azelastine, Fluticasone (Experimental): TEST = MP29-02 = Combination product Azelastine Hydrochloride and Fluticasone Propionate nasal spray (= US formulation as used in pivotal studies)
  Interventions: Drug: Azelastine, Fluticasone
- Fluticasone mono (Active Comparator): REF = FLU mono Fluticasone Propionate nasal spray (= essentially combination product formulation without any AZE; US FLU mono formulation as used in pivotal studies)
  Interventions: Drug: Fluticasone mono
- Fluticasone (Active Comparator): COMP = Fluticasone Propionate Nasal Spray, Roxane Laboratories = FLU mono Fluticasone propionate nasal spray (= US marketed product)
  Interventions: Drug: Fluticasone

INTERVENTIONS:
Drug: Azelastine, Fluticasone — TEST = MP29-02 = Combination product Azelastine Hydrochloride and Fluticasone Propionate nasal spray (= US formulation as used in pivotal studies)
  Arms: Azelastine, Fluticasone
Drug: Fluticasone mono — REF = FLU mono Fluticasone Propionate nasal spray (= essentially combination product formulation without any AZE; US FLU mono formulation as used in pivotal studies)
  Arms: Fluticasone mono
Drug: Fluticasone — COMP = Fluticasone Propionate Nasal Spray, Roxane Laboratories = FLU mono Fluticasone propionate nasal spray (= US marketed product)
  Arms: Fluticasone

SUMMARY:
The primary objective is to assess the effect of azelastine hydrochloride (AZE) on the relative bioavailability (AUC0-∞) of fluticasone propionate (FLU) when administered as fixed AZE-FLU combination product (TEST) compared to a similar formulation without containing AZE (i.e. FLU alone in the MP29-02 vehicle; REF).

The secondary objectives are to compare the relative bioavailability (AUC0-∞) of FLU when administered either as fixed AZE-FLU combination product (TEST) or as marketed FLU product, Fluticasone Propionate Nasal Spray, Roxane Laboratories (COMP); To compare the effects of AZE on other pharmacokinetic parameters of FLU (AUC0 tlast, CL/f, Cmax, tmax, t½); To assess adverse events.

DETAILED DESCRIPTION:
This study will enrol healthy subjects. It is considered that study results are more discriminative in healthy subjects than in rhinitis patients as there are no interferences by varying rhinitis symptoms and respective differences in the status of the nasal mucosa regarding the 3 study periods.

The time schedule for serum sampling (pre-dose and 8, 15, 30, 45 min, 1, 1¼, 1½, 2, 2½, 3, 4, 6, 8, 12, and 24 h p.a., time refer to the end of the second spray into the second nostril of each administration) is derived from previous bioavailability studies assuming a mean tmax of 1 h p.a. [P5] and a mean t1/2 of 3 h [L9]. Sampling times are expected to cover an AUC0-tlast above 80% of the total AUC of fluticasone propionate (bioanalytical detection method with a LLOQ of 0.5 pg/mL).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female healthy subjects of any Ethnic origin, age from 18 to 45 years.
2. Body mass index (BMI) from 18.5 to 30.0 kg/m2.
3. Use of adequate double contraception by female with childbearing potential (i.e. women of child bearing potential using a highly effective method of birth control defined as those which result in a low failure rate (i.e. <1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, hormonal IUDs) or surgically sterile (documented complete hysterectomy or bi-tubal ligations; partial hysterectomy is not sufficient or vasectomised partner). It must be ensured that the male partner uses a condom during intercourse (if not surgically sterilized).
4. Use of adequate double contraception by male, who is a sexually active man and has not been surgically sterilized, must consent that he uses a condom during intercourse and ensures that his female partner practices adequate contraception (a highly effective method of birth control defined as those which result in a low failure rate (i.e. <1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, hormonal IUDs) or surgically sterile (documented complete hysterectomy or bi-tubal ligations; partial hysterectomy is not sufficient).
5. Written informed consent.
6. Able to demonstrate correct nasal spray application technique at screening.

Exclusion Criteria:

1. History of allergic reaction or sensitivity to fluticasone propionate, azelastine hydrochloride or one of the excipients (e.g. benzalkoniumchloride, phenyl-ethyl alcohol, microcrystalline cellulose).
2. Any evidence of clinically relevant acute or chronic cardiovascular, pulmonary, hepatic, renal, gastrointestinal, haematological, endocrine, metabolic, mental, neurological, or other disease at screening.
3. Positive ß-HCG pregnancy test, or established pregnancy, breast-feeding or planned pregnancy during the study.

   Lack of suitability for the study:
4. History of haemophilia or coagulation disease.
5. Significant history of orthostatic hypotension, fainting or blackouts.
6. Existence of any surgical or medical condition, which might significantly alter the absorption, distribution, metabolism, or excretion of study drug.
7. Chronic or clinically relevant acute infections (e.g. of the respiratory tract including sinusitis and rhinitis), acute rhinorrhoea or febrile disease the week before randomisation.
8. Clinical chemical, haematological or any other laboratory parameters clinically relevant outside the reference range (e.g. elevated liver enzymes, renal laboratory parameters, and coagulation abnormalities such as abnormalities of platelet count, prothrombin time, or activated partial thromboplastin time).
9. Positive results in HIV, HCV and HBsAg tests.
10. ECG abnormalities of clinical relevance, in particular abnormal prolongations of QT/QTc- or PQ-interval (i.e. QTc according to Fridericia ≥ 450 ms, PQ ≥ 220 ms).
11. Resting heart rate in the awake subject below 45 BPM or above 90 BPM, systolic blood pressure below 100 mmHg or above 145 mmHg, diastolic blood pressure above 95 mmHg.
12. Regular therapy with corticosteroids (e.g. fluticasone propionate) or antihistamines (e.g. azelastine hydrochloride).
13. Any concurrent medication or any medication within 2 weeks preceding the start of the study (single intake/use of drugs may be accepted, if judged by the investigator to have no clinical relevance and no influence on study outcome).
14. Exposure to any cytochrome P450 3A4 inhibiting or inducing drug (e.g. ritonavir, ketoconazole, itraconazole, erythromycin, rifampicin, St. John's wort (Hypericum perforatum) etc.) diets (charcoal grilled meat, brussels sprouts, broccoli) or beverages (e.g. grapefruit juice) within 14 days prior to study enrolment, or anticipated consumption of such products during that period or at any time throughout the study.
15. History of any nasal surgery or known clinically relevant abnormalities, such as rhinitis medicamentosa, polyposis, septum deviation with clinical symptoms, or nasal structural abnormalities.
16. Known perennial airway allergies or vasomotor rhinitis. Known seasonal airway allergies which are clinically relevant acute within the last six weeks prior to the start of the study or might become acute during the study period.
17. History of malignancy within the past five years.
18. Blood donation within the last 2 months prior to the start of the study.
19. Present or history of drug or alcohol abuse within the last three years. Regular daily consumption of more than half a litre of usual beer or 0.25 L of wine per day or the equivalent quantity of approximately 30 g of alcohol in another form.
20. Current smoker or smoking during the last year.
21. Exposure to an investigational medicinal product within the last 3 months.
22. Subject reports a regular xanthine consumption of > 5 cups of coffee or black tea per day (or equivalent xanthine consumption of ≥ 500 mg xanthine per day using other products).
23. Subject is vegetarian or reports other strict dietary habits which would preclude the subject's acceptance of standardized meals.

    Administrative reasons:
24. Lack of ability or willingness to give informed consent.
25. Lack of willingness to have personal study related data collected, archived or transmitted according to protocol.
26. Lack of willingness or inability to co-operate adequately.
27. Anticipated non-availability for study visits/procedures.
28. Vulnerable subjects (such as persons kept in detention).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Effect of azelastine hydrochloride on the relative bioavailability of fluticasone | up to 24 h post application
  Effect of azelastine hydrochloride (AZE) on the relative bioavailability (AUC0-∞) of fluticasone propionate (FLU) when administered as fixed AZE-FLU combination product (TEST) compared to a similar formulation without containing AZE (i.e. FLU alone in the MP29-02 vehicle; REF).

SECONDARY OUTCOMES:
Relative bioavailability | up to 24 h post application
  Relative bioavailability (AUC0-∞) of FLU when administered either as fixed AZE-FLU combination product (TEST) or as marketed FLU product, Fluticasone Propionate Nasal Spray, Roxane Laboratories (COMP)
Effects of AZE on other pharmacokinetic parameters | up to 24 h post application
  Effects of AZE on other pharmacokinetic parameters of FLU (AUC0 tlast, CL/f, Cmax, tmax, t½)
Adverse Events | At and between treatment periods
  Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Christine Kolb, Study Director — MEDA Pharma GmbH & Co. KG
Locations (1):
- ClinPharmCologne, Cologne, North Rhine-Westphalia, Germany